CLINICAL TRIAL: NCT03856814
Title: Market Penetration of Laser Therapy in Venous Surgery: ZOL - ZMK Center Experience
Brief Title: Market Penetration of Laser Therapy in Venous Surgery: Ziekenhuis Oost-Limburg - Ziekenhuis Maas En Kempen Center Experience
Status: Completed | Type: Observational
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: BM-VL-01 ZOL
Record Dates: First submitted 2019-02-04; First posted 2019-02-27 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with varicose veins: Patients with varicose veins, indicative for treatment with EndoVenous Laser Ablation (EVLA) using the ELVeS® Radial® 2ring slim fiber or Surgery (ligation/stripping) according to the standard of care of the participating investigators.
  Interventions: Device: ELVeS® Radial® 2ring slim fiber used for EndoVenous Laser Ablation

INTERVENTIONS:
Device: ELVeS® Radial® 2ring slim fiber used for EndoVenous Laser Ablation — Device for endovenous laser ablation manufactured by Biolitec AG company (ELVeS system) - diode laser with a wavelength of 1470 nm

SUMMARY:
The goal of this registry is to evaluate the indication for EndoVenous Laser Ablation (EVLA) therapy. Can this be enhanced? What are the reasons for not using the laser? Therefore, this study aims to define clear indications for EVLA by registering the incentives of the participating investigators to use the laser instead of conventional corrective surgery for the treatment of varicose veins, at baseline and post-operative. Additionally, the efficacy and safety of the different varicose vein treatments will be evaluated by registering procedural characteristics, anatomic outcome (duplex ultrasound), quality of life (AVVQ) and postoperative pain (VAS).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old.
2. Patient must sign and date the informed consent form prior to treatment.
3. Presence of unilateral or bilateral primary or recurrent symptomatic varicose veins (CEAP grade ≥ C2).
4. Patient has an insufficient Great Saphenous Vein (GSV), Anterior Accessory Saphenous Vein (AASV) and/or Small Saphenous Vein (SSV), with venous symptoms (valve incompetence).

Exclusion Criteria:

1. Current deep vein thrombosis.
2. Acute superficial thrombosis.
3. Pregnancy.
4. Coagulopathy or bleeding disorders.
5. Contraindications to the use of general or regional anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients with varicose veins, indicative for treatment with Endovenous laser ablation (EVLA) or Surgery (ligation/stripping) according to routine patient care.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
To define clear indications for EndoVenous Laser Ablation (EVLA) treatment of varicose veins. | At baseline
  The participating investigators will register the incentives (based on clinical examination and/or anatomic outcome by duplex ultrasound, as well as secondary considerations) to use laser ablation or conventional treatment for varicose veins in the study database in order to define clear indications for EndoVenous Laser Ablation (EVLA) treatment of varicose veins and to investigate whether the use of EVLA can be enlarged.
To define clear indications for EndoVenous Laser Ablation (EVLA) treatment of varicose veins. | At 6 weeks follow-up
  The participating investigators will re-evaluate the chosen treatment option and document this re-evaluation in the study database in order to define clear indications for EndoVenous Laser Ablation (EVLA) treatment of varicose veins and to investigate whether the use of EVLA can be enlarged.

SECONDARY OUTCOMES:
Procedural characteristics | At index-procedure
  Type of anesthesia
Procedural characteristics | At index-procedure
  Number, type and length of veins treated
Procedural characteristics | At index-procedure
  Total energy per patient and fiber (when using the ELVeS® Radial® 2ring slim fiber)
Procedural characteristics | At index-procedure
  Number of procedures showing technical success, defined as the ability to treat the varicose veins as planned
Procedural characteristics | At index-procedure
  Peri-operative adverse events (bleeding, incomplete treatment, technical defects, difficult visualization, …)
Procedural characteristics | At index-procedure
  Duration of the index-procedure
Pain scoring using the Visual Analog Scale (VAS) | At discharge, up to 1 week
  The VAS scale contains a 0 - 100 grading with 0 equaling no pain and 100 equaling the worst conceivable pain. The patient is asked to select the number on the scale that corresponds to the worst level of pain he/she experiences. Pain is classified into mild (1 - 30 mm), moderate (31 - 60 mm) and severe (61 - 100 mm). Absence of pain is defined as VAS = 0.
Pain scoring using the Visual Analog Scale (VAS) | At 6 weeks follow-up
  The VAS scale contains a 0 - 100 grading with 0 equaling no pain and 100 equaling the worst conceivable pain. The patient is asked to select the number on the scale that corresponds to the worst level of pain he/she experiences. Pain is classified into mild (1 - 30 mm), moderate (31 - 60 mm) and severe (61 - 100 mm). Absence of pain is defined as VAS = 0.
Anatomic success of EndoVenous Laser Ablation (EVLA) | At 6 weeks follow-up
  Defined as occlusion of the treated veins and lack of reflux objectified with duplex ultrasonography.
Quality of life by scoring Aberdeen Varicose Vein Questionnaire (AVVQ) | At baseline
  Aberdeen Varicose Vein Questionnaire (AVVQ) is a validated tool for assessing the perceived health of patients with varicose veins. The AVVQ comprises 13 quality of life questions, including a set of manikin legs, on which participants are asked to draw their veins.
Quality of life by scoring Aberdeen Varicose Vein Questionnaire (AVVQ) | At 6 weeks follow-up
  Aberdeen Varicose Vein Questionnaire (AVVQ) is a validated tool for assessing the perceived health of patients with varicose veins. The AVVQ comprises 13 quality of life questions, including a set of manikin legs, on which participants are asked to draw their veins.
Quality of life by scoring Aberdeen Varicose Vein Questionnaire (AVVQ) | At 6 months follow-up
  Aberdeen Varicose Vein Questionnaire (AVVQ) is a validated tool for assessing the perceived health of patients with varicose veins. The AVVQ comprises 13 quality of life questions, including a set of manikin legs, on which participants are asked to draw their veins.
Post-operative adverse events | At discharge, up to 1 week
  Number of participants with numbness, persistent bruising, skin loss or ulceration, hematoma, infection, bleeding, deep venous thrombosis, etc.
Post-operative adverse events | At 6 weeks follow-up
  Number of participants with numbness, persistent bruising, skin loss or ulceration, hematoma, infection, bleeding, deep venous thrombosis, etc.
Post-operative adverse events | At 6 months follow-up
  Number of participants with numbness, persistent bruising, skin loss or ulceration, hematoma, infection, bleeding, deep venous thrombosis, etc.
Re-interventions | At discharge, up to 1 week
  Number of participants with re-interventions
Re-interventions | At 6 weeks follow-up
  Number of participants with re-interventions
Re-interventions | At 6 months follow-up
  Number of participants with re-interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg (Sint-Jan,Genk; Sint-Barbara,Lanaken; ZMK,Maaseik), Genk, Limburg, Belgium